CLINICAL TRIAL: NCT04843540
Title: A Phase 1 Open-Label Study to Assess the Effect of a Strong CYP3A4 Inducer, Rifampin, on the Single Dose Pharmacokinetic Profile of CTP-543 in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of CTP-543 and Rifampin in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Concert Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CP543.1008
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers
Keywords: Rifampin; Drug-drug interaction; CTP-543

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTP-543 (Experimental): On Day 1, participants will receive a single oral dose of CTP-543. Following a washout period on Days 2 and 3, participants will receive a single oral dose of rifampin on Day 4 through Day 15, with a single oral dose of CTP-543 being co-administered on Day 14.
  Interventions: Drug: CTP-543

INTERVENTIONS:
Drug: CTP-543 — Rifampin as oral capsule

SUMMARY:
This is a Phase 1 open-label study of the effect of rifampin on the pharmacokinetics of CTP-543 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study
* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at Screening
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs
* If of reproductive age, willing and able to use a medically highly effective form of birth control 30 days prior to first dose, during the study and for 30 days following last dose of study medication
* Understands the study procedures in the informed consent form, and be willing and able to comply with the protocol

Exclusion Criteria:

* History or presence of clinically significant medical or psychiatric condition or disease
* History of any illness that might confound the results of the study or poses an additional risk to the subject by their participation in the study
* History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing
* Females who are nursing, pregnant, or planning to become pregnant while in the study, and for 30 days after last dose of study drug
* Positive results at Screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* A positive test or history of incompletely treated or untreated tuberculosis
* Donation of > 499 mL of blood or plasma within 56 days of Screening (during a clinical trial or at a blood bank donation) and for 30 days after last dose of study drug

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
AUC0-t | 16 hours
  Area Under the Plasma Concentration-Time Profile
AUC0-inf | 16 hours
  Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time
Cmax | 16 hours
  Maximum observed concentration of drug in plasma
Tmax | 16 hours
  Time to reach maximum observed concentration of drug in plasma

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 47 days
  An adverse event is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Pharmacology of Miami, Miami, Florida, United States